CLINICAL TRIAL: NCT04985773
Title: A Study to EXhibit Percutaneous Coronary Artery Dilatation With Non-Slip Element Balloon (EXPANSE-PTCA)
Brief Title: A Study to EXhibit Percutaneous Coronary Artery Dilatation With Non-Slip Element Balloon
Acronym: EXPANSE-PTCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Infraredx (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDX-CL-5000
Record Dates: First submitted 2021-07-21; First posted 2021-08-02 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Coronary Stenosis; Coronary Artery Stenosis; In-stent Restenosis
Keywords: Coronary dilation catheter; Percutaneous coronary artery dilatation; Non-slip Element balloon; Restenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Intervention Model Description: A prospective, multi-center, single arm clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Lacrosse NSE ALPHA percutaneous coronary intervention (PCI) (Experimental): Percutaneous coronary intervention (PCI) in which at least one Lacrosse NSE ALPHA device is used.
  Interventions: Device: Lacrosse NSE ALPHA coronary dilatation catheter

INTERVENTIONS:
Device: Lacrosse NSE ALPHA coronary dilatation catheter — The Lacrosse NSE ALPHA is a rapid exchange percutaneous transluminal coronary angioplasty balloon catheter with non-slip element nylon threads that focus dilatation force to reduce balloon slippage during inflation.

SUMMARY:
The objective of this study is to evaluate safety and effectiveness of the Lacrosse NSE ALPHA coronary dilatation catheter during PCI in subjects with stenotic coronary arteries.

DETAILED DESCRIPTION:
The investigation is a prospective, multi-center, single arm clinical study. The study will be conducted in up to 15 investigational sites in the U.S. This study will enroll and treat 200 subjects, including a minimum of 30 subjects with in-stent restenosis (ISR).

The population for this study is subjects with stenotic coronary artery disease who are suitable candidates for PTCA.

After screening for initial inclusion and exclusion criteria, eligible subjects will be asked to participate in the study by signing a consent form. Following consent, subjects will undergo a baseline visit where additional eligibility criteria will be assessed. An angiogram will be completed to assess for angiographic eligibility. If a non-target lesion is identified, it must be treated successfully prior to target lesion treatment. Once treatment of the target lesion(s) has been attempted, the subject will be considered enrolled in the study.

Subjects will be followed through hospital discharge.

ELIGIBILITY:
INCLUSION CRITERIA

General inclusion criteria:

1. Age 18 years or older.
2. Willing to provide written informed consent and written HIPAA authorization prior to initiation of study-related procedures.
3. Agree to not participate in any other clinical study during hospitalization for the index procedure that would interfere with the endpoints of this study.
4. Clinical evidence of ischemic heart disease, stable/unstable angina, or silent ischemia.
5. Acceptable candidate for PCI and emergency coronary artery bypass grafting and is planned for possible PTCA and/or stent placement.

   Angiographic inclusion criteria:
6. De novo or restenotic lesion(s) in native coronary arteries, including in-stent restenosis.
7. A maximum of two lesions, including at least one target lesion, in single or double vessel coronary artery disease.

   1. If two target lesions are defined, then no non-target lesions can be treated.
   2. If a single target lesion is defined, then a single non-target lesion may be treated, but if so, it must be located in a different coronary artery from the target lesion.
8. Target lesion(s) must have a reference vessel diameter between 2.0 mm and 4.0 mm by visual estimation.
9. Target lesion(s) must have a diameter stenosis of (a) ≥70% by visual estimation or (b) >50% by visual estimation and a fractional flow reserve (FFR) of <0.80 or resting full-cycle ratio (RFR) or instantaneous wave-free ratio (iFR) <0.9.
10. Treatment of non-target lesion, if any, must be completed prior to treatment of target lesion; must not, in the opinion of the investigator, impact the conduct or completion of the index procedure; and must be deemed a clinical angiographic success as visually assessed by the investigator.

EXLUSION CRITERIA

General exclusion criteria:

1. Known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, anti-platelet medications, a clopidogrel non-responder, or sensitivity to contrast media that cannot be adequately pre-medicated or replaced with a clinically suitable alternative.
2. Known diagnosis of type I myocardial infarction (resulting from primary reduction of flow from a culprit lesion likely to have a thrombotic component) within 7 days prior to the index procedure.
3. Known pregnancy or is nursing. Women of child-bearing potential should have a documented negative pregnancy test within 7 days prior to index procedure.
4. Planned target lesion treatment with atherectomy (rotational, orbital or laser), cutting balloon, thrombectomy, lithotripsy or an unapproved device during the index procedure.
5. Serum creatinine >2.0 mg/dl within 7 days prior to the index procedure.
6. Cerebrovascular accident within 6 months prior to the index procedure.
7. Active peptic ulcer or active gastrointestinal bleeding within 6 months prior to the index procedure.
8. Left ventricular ejection fraction <30% based on most recent measurement within a year of the index procedure (if LVEF is not available in the medical records, it may be obtained at the time of the index procedure, prior to enrollment).
9. Target lesion located within a bypass graft (venous or arterial) or graft anastomosis.
10. Previous percutaneous intervention, within 9 months before the study procedure, on lesions in a target vessel (including side branches) that are located within 10 mm from the current target lesion(s).
11. Target lesion(s) with complete total occlusion defined as the complete obstruction of a native coronary artery, exhibiting TIMI 0 or TIMI 1 flow, with an occlusion duration of at least 3 months.
12. Unstable hemodynamics or shock.
13. Other medical condition which might, in the opinion of the investigator, put the patient at risk or confound the results of the study.

    Angiographic exclusion criteria
14. Target lesion(s) longer than 32 mm by visual estimation.
15. Extreme angulation (90º or greater) within 5 mm of the target lesion.
16. Target lesion(s) demonstrating flow limiting dissection (NHLBI Grade C or higher) prior to deployment of the Lacrosse NSE ALPHA.
17. Unprotected left main coronary artery disease (>50% diameter stenosis).
18. Coronary artery spasm of the target vessel in the absence of a significant stenosis.
19. Target lesion(s) with angiographic presence of probable or definite thrombus.
20. Target lesion(s) involves a bifurcation requiring treatment with more than one stent or pre-dilatation of a side branch >2.0 mm in diameter.
21. Target lesion(s) located in bifurcation beyond stent struts.
22. Target lesion(s) located distal to an implanted stent.
23. Target lesion(s) with stent damage.
24. Non-target lesion that meets any of the following criteria:

    * Located within a bypass graft (venous or arterial)
    * Located in an unprotected left main coronary artery
    * A CTO
    * Involves a bifurcation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Krucoff, MD, Principal Investigator — Duke University
Locations (10):
- United States (10):
  - VA Palo Alto Health System, Palo Alto, California
  - Baptist Health Lexington, Lexington, Kentucky
  - M Health Fairview, Maplewood, Minnesota
  - Minneapolis Heart Institute - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Cardiology Associates Research, Tupelo, Mississippi
  - Columbia University Medical Center, New York, New York
  - Cornell University, New York, New York
  - St Francis Hospital, Roslyn, New York
  - Ascension Saint Thomas Heart West, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI)
Started | 200
Completed | 199
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI)
Number analyzed (Participants) | 200
Age, Continuous [Median (Full Range); unit: years] | 69.5 [32.0 to 93.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 157
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 171
  Other | 10
  Black or African American | 8
  Subject chose not to disclose | 7
  Asian | 3
  American Indian or Alaska Native | 1
Region of Enrollment [Number; unit: participants]
  United States | 200

OUTCOME MEASURES:

1. Primary Outcome: Procedure Success
Description: Defined as:
  * Successful delivery, inflation, deflation, and withdrawal of the study balloon; and
  * No evidence of device-related vessel perforation, flow limiting dissection (grade C or higher per Clinical Events Committee (CEC) adjudication) or reduction in thrombolysis in myocardial infarction (TIMI) flow from baseline (per core laboratory assessment); and
  * Final TIMI flow grade of 3 at the conclusion of the PCI procedure per core laboratory assessment.
  This endpoint will be presented as the proportion of subjects experiencing device procedural success.
Time Frame: Procedural
Population: Four (4) subjects had no final TIMI assessed by either the core lab or the site so are not included in the assessment of primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI)
Number analyzed (Participants) | 196
Participants | 176

2. Secondary Outcome: Percentage of Subjects With Angiographic Procedural Success
Description: Defined as final diameter stenosis ≤50% in at least one of the Lacrosse NSE ALPHA attempted lesions following completion of the interventional procedure, including adjunctive stenting per core lab assessment.
Time Frame: Procedural
Population: Three (3) subjects were missing final diameter stenosis (both core lab and site data).
Measure: Count of Participants; unit: Participants
Arm/Group | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI)
Number analyzed (Participants) | 197
Participants | 197

3. Secondary Outcome: Percentage of Subjects With a MACE
Description: Defined as a composite of:
  * All-cause death
  * Myocardial infarction (MI)
  * Clinically indicated target lesion revascularization (TLR)
Time Frame: At hospital discharge, an average of 1 day after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI)
Number analyzed (Participants) | 200
Participants | 1

4. Secondary Outcome: Percentage of Subjects With Stent Thrombosis Within the Target Vessel(s)
Description: Stent thrombosis is defined using ARC-2 definitions for definite & probable per CEC adjudication.
Time Frame: At hospital discharge, an average of 1 day after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI)
Number analyzed (Participants) | 200
Participants | 0

5. Secondary Outcome: Percentage of Subjects With a Clinically Significant Arrhythmia
Description: A clinically significant arrhythmia is defined as those requiring intervention.
Time Frame: At hospital discharge, an average of 1 day after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI)
Number analyzed (Participants) | 200
Participants | 4

6. Secondary Outcome: Occurrence of Lacrosse NSE ALPHA Balloon Rupture
Description: Per device deficiency eCRF
Time Frame: Procedural
Measure: Count of Participants; unit: Participants
Arm/Group | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI)
Number analyzed (Participants) | 200
Participants | 1

7. Secondary Outcome: Change in Minimum Lumen Diameter (MLD) Following Use of the Lacrosse NSE ALPHA Catheter
Description: Measured by quantitative coronary angiography (QCA). A positive value represents an increase in MLD compared to baseline. A negative value represents a decrease in MLD compared to baseline.
Time Frame: Procedural
Population: Only subjects that had lesions were analyzed (N=147). If final diameter stenosis or MLD was not assessed by the core laboratory, due to missing imaging, site-reported data was used, if available.
Measure: Median (Full Range); unit: mm
Units Other Than Participants: lesions
Arm/Group | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI)
Number analyzed (Participants) | 147
Number analyzed (lesions) | 158
mm | 0.7 [0.1 to 2.2]

8. Secondary Outcome: Device Procedural Success (Per Target Lesion)
Description: Successful delivery, inflation, deflation, and withdrawal of the study balloon; and no evidence of device-related vessel perforation, flow limiting dissection (grade C or higher) or reduction in thrombolysis in myocardial infarction (TIMI) flow from baseline; and final TIMI flow grade of 3 at the conclusion of the PCI procedure. This endpoint will be presented as the proportion of target lesions experiencing device procedural success.
Time Frame: Procedural
Population: Includes only those lesions in the subjects included in the primary endpoint analysis; four (4) subjects had no final TIMI assessed by either the core lab or the site so are not included in the assessment of primary endpoint.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI)
Number analyzed (Participants) | 196
Number analyzed (lesions) | 216
lesions | 193

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the point of subject enrollment through study completion at hospital discharge (hospital stay expected to be an average of 24 hours).
Arm/Group | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI)
All-Cause Mortality (participants affected / at risk) | 1/200
Serious Adverse Events (participants affected / at risk) | 20/200
Other Adverse Events (participants affected / at risk) | 17/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI) (N=200)
Myocardial infarction (Cardiac disorders) | 1 (1)
Arterial dissection (Vascular disorders) | 4 (4)
Hematoma, access site, >5 cm (Injury, poisoning and procedural complications) | 2 (2)
Blood loss from puncture site (General disorders) | 2 (2)
Chest pain, non-cardiac (General disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Arrhythmia, bradycardia (Cardiac disorders) | 2 (2)
Arrhythmia, other (Cardiac disorders) | 1 (1)
Arterial perforation (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Other, chest pain (General disorders) | 1 (1)
Arterial occlusion of the second diagonal (Vascular disorders) | 1 (1)
Hematamesis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lacrosse NSE ALPHA Percutaneous Coronary Intervention (PCI) (N=200)
Arterial dissection (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT04985773/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT04985773/SAP_001.pdf